CLINICAL TRIAL: NCT06305234
Title: A Multi-Center, Prospective, Longitudinal, Study Evaluating Immunologic, Inflammatory, and Laboratory Parameters Associated With Long-Term Palynziq® (Pegvaliase) Treatment in Subjects With Phenylketonuria (PKU) in the United States
Brief Title: A Long Term, Post-marketing Study of Immune Response in Patients Receiving Palynziq Treatment for PKU (PALisade)
Status: Recruiting | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 165-503
Record Dates: First submitted 2024-01-30; First posted 2024-03-12 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Phenylketonuria (PKU)
Keywords: PKU; Phenylketonuria; Palynziq; pegvaliase; observational; safety study; immunogenicity assessment; inflammatory assessment
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A small blood sample may be kept to be used only in a health authority request.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Pegvaliase — Must be enrolled in the 165-501 PALace study. Subjects currently receiving or who plan to receive pegvaliase treatment within 30 days after the date of enrollment in the 165-501 study, including subjects who previously received pegvaliase as part of the clinical development program and have completed study participation

SUMMARY:
This is a 10-year multi-center, prospective, longitudinal, single arm study evaluating immunologic, inflammatory and laboratory parameters associated with long-term Palynziq treatment in subjects with phenylketonuria (PKU) in the United States (US). Subjects in the US for whom a clinical decision has been made that they will receive pegvaliase to treat their PKU within 30 days following the date of enrollment in Study 165-501 (incident-users) or who have previously started treatment with pegvaliase at the date of enrollment in Study 165-501 (prevalent-users) are eligible for participation in Study 165-503.

DETAILED DESCRIPTION:
This is a 10-year multi-center, prospective, longitudinal, single arm study evaluating immunologic, inflammatory and laboratory parameters associated with long-term Palynziq treatment in subjects with phenylketonuria (PKU) in the United States (US). Subjects in the US for whom a clinical decision has been made that they will receive pegvaliase to treat their PKU within 30 days following the date of enrollment in Study 165-501 (incident-users) or who have previously started treatment with pegvaliase at the date of enrollment in Study 165-501 (prevalent-users) are eligible for participation in Study 165-503. Subjects participating in the 165-501 study who consent to participate in this study (165-503) will be requested to provide pre-dose blood samples for Phe, immunologic and inflammatory marker testing approximately every 3 months for the first 3 years of participation, then every 6 months for the remainder of the study. Subjects will be requested to provide additional pre-dose blood samples at the time of Study 165-501 -protocol defined safety events. Additional pre-dose samples will be drawn as per standard of care as detailed in protocol 165-501. The blood Phe, immunologic (PAL IgG, PEG IgG, PEG IgM, anti-pegvaliase IgE), and inflammatory (C3/C4, hsCRP) markers, will be sent to a central laboratory for processing. Data collected in the 165-501 study will be combined with the data collected in this study to decrease burden on sites for data entry and to avoid duplication of ADR reporting (see Criteria for Evaluation). The combined data will be reported in the Clinical Study Report for this study. Subjects can withdraw from Study 165-503 and remain on Study 165-501, but they cannot withdraw from Study 165-501 and remain on Study 165-503 as safety events and other data-points are collected in Study 165-501.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled at US sites participating in the 165-501 study.

Exclusion Criteria:

* Legal incapacity or limited legal capacity without legal guardian representation.
* Subject is unable or unwilling to provide informed consent for the additional interventional burden of the study (blood sampling).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects enrolled at US sites participating in the 165-501 study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2033-11-18 (Estimated); Study Completion 2033-11-18 (Estimated)

PRIMARY OUTCOMES:
To evaluate immunologic and inflammatory responses associated with occurrences of | A maximum of 10 years treatment duration.
  * Acute systemic hypersensitivity reaction
  * Anaphylaxis
  * Angioedema
  * Serum sickness
  * Severe hypersensitivity reaction
  * Severe or Persistent arthralgia
  * Severe injection site reaction

SECONDARY OUTCOMES:
Evaluation of immunologic and/or inflammatory responses over time | A maximum of 10 years treatment duration.
  To evaluate immunologic and inflammatory responses (immunologic testing, inflammatory markers) associated with occurrences of end-organ function (eg, kidney, liver) related, immune-mediated adverse drug reactions (ADRs)*
Evaluation of immunologic responses over time | A maximum of 10 years treatment duration.
  To evaluate the potential association between immunologic responses and blood Phe levels
  * A list of end-organ function related, immune-mediated ADRs is included as an appendix to the statistical analysis plan (SAP).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (6):
- United States (6):
  - University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas